CLINICAL TRIAL: NCT04593043
Title: Replication of the RELY Anticoagulant Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-RELY
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Warfarin; Dabigatran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Warfarin: Reference group
  Interventions: Drug: Warfarin
- Dabigatran: Exposure group
  Interventions: Drug: Dabigatran

INTERVENTIONS:
Drug: Warfarin — Warfarin dispensing claim is used as the reference
  Groups: Warfarin
Drug: Dabigatran — Dabigatran dispensing claim is used as the exposure
  Groups: Dabigatran

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Please see: https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Eligible cohort entry dates: Market availability of dabigatran in the U.S. started on October 19, 2010. For Marketscan: Oct 19, 2010 -Dec 31, 2018 (end of data availability). For Optum: Oct 19, 2010 -Dec 31, 2019 (end of data availability). For Medicare: Oct 19, 2010 -Dec 31, 2017.

Inclusion Criteria:

* 1. AF documented as follows: (1a or 1b or 1c)

  * 1a. There is ECG documented AF on the day of screening or randomization
  * 1b. The patient has had a symptomatic episode of paroxysmal or persistent AF documented by 12-lead ECG within 6 m before randomization
  * 1c. There is documentation of symptomatic or asymptomatic paroxysmal or persistent AF on 2 separate occasions, at least 1 day apart, one of which is within 6 m before randomization.
* 2. In addition to documented AF, patients must have one of the following: (2a or 2b or 2c or 2d or 2e)

  * 2a. History of previous stroke, TIA, or systemic embolism
  * 2b. Ejection fraction <40% documented by echocardiogram, radionuclide or contrast angiogram in the last 6 m
  * 2c. Symptomatic heart failure, New York Heart Association class 2 or higher in the last 6 m
  * 2d. Age ≥75 y
  * 2e. Age ≥65 y and one of the following:

    * Diabetes mellitus on treatment
    * Documented coronary artery disease (any of: prior myocardial infarction, positive stress test, positive nuclear perfusion study, prior CABG surgery or PCI, angiogram showing ≥75% stenosis in a major coronary artery
    * Hypertension requiring medical treatment
* 3. Age >18 y at entry

Exclusion Criteria:

* 1. History of heart valve disorders (ie, prosthetic valve or hemodynamically relevant valve disease)
* 2. Severe, disabling stroke within the previous 6 months or Any stroke within the previous 14 days
* 3. Conditions associated with an increased risk of bleeding:

  * 3a. Major surgery in the previous month
  * 3c. History of intracranial, intraocular, spinal, retroperitoneal or atraumatic intra-articular bleeding
  * 3d. Gastrointestinal hemorrhage within the past year
  * 3e. Symptomatic or endoscopically documented gastroduodenal ulcer disease in the previous 30 days
  * 3f. Hemorrhagic disorder or bleeding diathesis
  * 3i. Uncontrolled hypertension (systolic blood pressure >180 mm Hg and/ or diastolic blood pressure >100 mm Hg)
* 7. Severe renal impairment (estimated creatinine clearance ≤30 mL/min)
* 8. Active infective endocarditis
* 9. Active liver disease
* 10. Women who are pregnant or of childbearing potential who refuse to use a medically acceptable form of contraception throughout the study
* 11. Anemia (hemoglobin level < 100g/L) or thrombocytopenia (platelet count <100 × 109/L)
* 14. Patients considered unreliable by the investigator or have a life expectancy less than the expected duration of the trial because of concomitant disease, or has any condition which in the opinion of the investigator, would not allow safe participation in the study (eg, drug addiction, alcohol abuse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, cohort study design comparing dabigatran to warfarin. The patients will be required to have continuous enrollment during baseline period of 180 days before initiation of dabigatran or the comparator drug (cohort entry date). Follow-up for the outcome, begins the day after drug initiation.
Sampling Method: Probability Sample
Enrollment: 78140 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Relative hazard of composite outcome of Stroke and Systemic Embolism | [Time Frame: Through study completion (a median of 98 days)]
  Relative hazard of composite outcome of Stroke and Systemic Embolism - Please refer to uploaded protocol for full definition due to size limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham And Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT04593043/Prot_SAP_002.pdf